CLINICAL TRIAL: NCT00592553
Title: A Phase 2B Efficacy and Safety Study of PTC124 in Subjects With Nonsense-Mutation-Mediated Duchenne and Becker Muscular Dystrophy
Brief Title: Phase 2B Study of PTC124 (Ataluren) in Duchenne/Becker Muscular Dystrophy (DMD/BMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-007-DMD; 2007-005478-29 (EudraCT Number)
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Becker muscular dystrophy; Nonsense mutation; Premature stop codon; DMD/BMD; PTC124
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-Dose Ataluren (Experimental): Participants will receive ataluren suspension orally 3 times a day (TID), 20 milligrams/kilogram (mg/kg) at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for 48 weeks.
  Interventions: Drug: Ataluren
- Low-Dose Ataluren (Experimental): Participants will receive ataluren suspension orally TID, 10 mg/kg at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 48 weeks.
  Interventions: Drug: Ataluren
- Placebo (Placebo Comparator): Participants will receive placebo matched to ataluren orally TID at morning, midday, and evening for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the respective arms.
  Other Names: PTC124
  Arms: High-Dose Ataluren; Low-Dose Ataluren
Drug: Placebo — Placebo matching to ataluren will be administered as the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
DMD/BMD is a genetic disorder that develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability during childhood and teenage years. A specific type of mutation, called a nonsense (premature stop codon) mutation is the cause of DMD/BMD in approximately 13 percent (%) of boys with the disease. Ataluren is an orally delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 2b trial that will evaluate the clinical benefit of ataluren in boys with DMD/BMD due to a nonsense mutation. The main goals of the study are to understand whether ataluren can improve walking, activity, muscle function, and strength and whether the drug can safely be given for a long period of time.

DETAILED DESCRIPTION:
This study is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, dose-ranging, efficacy and safety study, designed to document the clinical benefit of ataluren when administered as therapy of patients with DMD/BMD due to a nonsense mutation (premature stop codon) in the dystrophin gene.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if <18 years of age).
* Male sex.
* Age ≥5 years.
* Phenotypic evidence of DMD/BMD based on the onset of characteristic clinical symptoms or signs (that is, proximal muscle weakness, waddling gait, and Gowers' maneuver) by 9 years of age, an elevated serum CK level, and ongoing difficulty with ambulation.
* Documentation of the presence of a nonsense point mutation in the dystrophin gene as determined by gene sequencing from a laboratory certified by the College of American Pathologists (CAP), the Clinical Laboratory Improvement Act/Amendment (CLIA), or an equivalent organization.
* Documentation that a blood sample has been drawn for confirmation of the presence of a nonsense mutation in the dystrophin gene.
* Ability to walk ≥75 meters unassisted during the screening 6-minute walk test. Note: Other personal assistance or use of assistive devices for ambulation (for example, short leg braces, long leg braces or walkers) were not permitted.
* Confirmed screening laboratory values within the central laboratory ranges (hepatic, adrenal, renal, and serum electrolytes parameters).
* In participants who were sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and 6-week follow-up periods.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions. Note: Psychological, social, familial, or geographical factors that might preclude adequate study participation (in particular, the ability to satisfactorily perform the 6MWT) should have been considered.

Exclusion Criteria:

* Treatment with systemic aminoglycoside antibiotics within 3 months prior to start of study treatment.
* Initiation of systemic corticosteroid therapy within 6 months prior to start of study treatment or change in systemic corticosteroid therapy (for example, initiation, change in type of drug, dose modification not related to body weight change, schedule modification, interruption, discontinuation, or reinitiation) within 3 months prior to start of study treatment.
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or reinitiation) in prophylaxis/treatment for congestive heart failure within 3 months prior to start of study treatment.
* Treatment with warfarin within 1 month prior to start of study treatment.
* Prior therapy with ataluren.
* Known hypersensitivity to any of the ingredients or excipients of the study drug (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab-O-Sil® M5P [colloidal silica], magnesium stearate).
* Exposure to another investigational drug within 2 months prior to start of study treatment.
* History of major surgical procedure within 30 days prior to start of study treatment.
* Ongoing immunosuppressive therapy (other than corticosteroids).
* Ongoing participation in any other therapeutic clinical trial.
* Expectation of major surgical procedure (for example, scoliosis surgery) during the 12-month treatment period of the study.
* Requirement for daytime ventilator assistance.
* Clinical symptoms and signs of congestive heart failure (American College of Cardiology/American Heart Association Stage C or Stage D) or evidence on echocardiogram of clinically significant myopathy.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, electrocardiogram findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Consistent with the X-linked genetic basis and natural history of DBMD, all of the participants were males.
Enrollment: 174 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leone Atkinson, MD, PhD, Study Director — PTC Therapeutics
Locations (37):
- United States (15):
  - University of California-Davis, Sacramento, California
  - The Children's Hospital, Aurora, Colorado
  - Child Neurology Center of Pensacola, Pensacola, Florida
  - University of Iowa Healthcare, Iowa City, Iowa
  - University of Kansas Medical Centre, Kansas City, Kansas
  - Children's Hospital of Boston/Harvard Medical School, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical School, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Southwestern University, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Institute For Neuromuscular Research, The Children's Hospital at Westmead, Westmead
- University Hospital KU Leuven, Leuven, Belgium
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
- France (3):
  - Service de Neuropediatrie, hôpital La Timone, Marseille
  - Neuromuscular center of Nantes, Nantes
  - Groupe Hospitalier La Pitie-Salpetriere, Paris
- Germany (2):
  - University Clinic for Children, University of Essen, Essen
  - University Hospital, Freiburg im Breisgau
- Hadassah Medical Center, Hebrew University Hospital, Jerusalem, Israel
- Italy (3):
  - Ospedale Maggiore Policlinico in Milan, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
  - U.O. Complessa di Neuropsichiatria Infantile, Rome
- Spain (2):
  - Hospital Sant Joan de déu, Barcelona
  - Hospital Universitari La Fe, Valencia
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Pediatric Hospital, Stockholm
- United Kingdom (3):
  - Imperial College London, Hammersmith Hospital, London
  - Univ of Newcastle, Institute of Human Genetics, Newcastle
  - Robert Jones and Agnes Hunt Orthopaedic NHS Trust, Oswestry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei YS, Hnaini M, ElAloul B, Zapata E, Campbell C. Duchenne Muscular Dystrophy Fatigue Trajectories. Neuropediatrics. 2024 Feb;55(1):42-48. doi: 10.1055/a-2101-7860. Epub 2023 May 26. PMID 37236246
- [Derived] Shieh PB, Elfring G, Trifillis P, Santos C, Peltz SW, Parsons JA, Apkon S, Darras BT, Campbell C, McDonald CM; Members of the Ataluren Phase IIb Study Group; Members of the Ataluren Phase IIb Study Clinical Evaluator Training Group; Members of the ACT DMD Study Group; Members of the ACT DMD Clinical Evaluator Training Group. Meta-analyses of deflazacort versus prednisone/prednisolone in patients with nonsense mutation Duchenne muscular dystrophy. J Comp Eff Res. 2021 Dec;10(18):1337-1347. doi: 10.2217/cer-2021-0018. Epub 2021 Oct 25. PMID 34693725
- [Derived] Campbell C, Barohn RJ, Bertini E, Chabrol B, Comi GP, Darras BT, Finkel RS, Flanigan KM, Goemans N, Iannaccone ST, Jones KJ, Kirschner J, Mah JK, Mathews KD, McDonald CM, Mercuri E, Nevo Y, Pereon Y, Renfroe JB, Ryan MM, Sampson JB, Schara U, Sejersen T, Selby K, Tulinius M, Vilchez JJ, Voit T, Wei LJ, Wong BL, Elfring G, Souza M, McIntosh J, Trifillis P, Peltz SW, Muntoni F; PTC124-GD-007-DMD Study Group; ACT DMD Study Group; Clinical Evaluator Training Groups. Meta-analyses of ataluren randomized controlled trials in nonsense mutation Duchenne muscular dystrophy. J Comp Eff Res. 2020 Oct;9(14):973-984. doi: 10.2217/cer-2020-0095. Epub 2020 Aug 27. PMID 32851872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 185 participants were screened for eligibility, of which 11 participants did not meet entry criteria.
Pre-assignment Details: A total of 174 eligible participants were randomized in 1:1:1 ratio to receive either placebo, low-dose ataluren, or high-dose ataluren.
Groups:
- High-Dose Ataluren: Participants received ataluren suspension orally 3 times a day (TID), 20 milligrams/kilogram (mg/kg) at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for 48 weeks.
- Low-Dose Ataluren: Participants received ataluren suspension orally TID, 10 mg/kg at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for 48 weeks.
- Placebo: Participants received placebo matched to ataluren orally TID at morning, midday, and evening for 48 weeks.
Period: Overall Study
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Started | 60 | 57 | 57
As-treated Population (All Randomized participants who received any study treatment.) | 60 | 57 | 57
ITT Population (Received any study treatment; had a valid baseline, and at least 1 valid post-baseline 6MWD value.) | 60 | 57 | 57
Completed | 59 | 57 | 57
Not Completed | 1 | 0 | 0
Not completed — Protocol Noncompliance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all randomized participants who actually received any study treatment.
Groups:
- High-Dose Ataluren: Participants received ataluren suspension orally TID, 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo | Total
Number analyzed (Participants) | 60 | 57 | 57 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (2.53) | 8.8 (2.91) | 8.3 (2.33) | 8.5 (2.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 60 | 57 | 57 | 174
6-Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] — The 6MWD test was performed in a 30-meters-long flat corridor, where the participant was instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
  meters | 358.2 (103.97) | 350.0 (97.55) | 359.6 (87.67) | 356.0 (96.30)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6MWD at Week 48
Description: The 6MWD test was performed in a 30 meters long flat corridor, where the participant was instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
Time Frame: Baseline, Week 48
Population: Intent-to-treat (ITT) population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 59 | 55 | 55
meters | -41.81 (89.234) | -12.86 (72.007) | -42.56 (90.046)
Statistical Analysis 1: Comparison: High-Dose Ataluren vs Placebo; Analysis was performed using mixed model for repeated measures (MMRM) method including rank transformed 6MWD as the dependent variable; and rank transformed baseline 6MWD, treatment, visit, age (less than [<] 9 years versus [vs.] greater than or equal to [>=] 9 years) and corticosteroid use (yes vs. no) stratification factors, and interaction between treatment and visit as independent variables; Test type: Other; p = 0.4756, Mixed Models Analysis; Least Square (LS) Mean Difference = -30.52, 95% CI 2-sided [-114.8 to 53.75], Standard Error of Mean 42.68
Statistical Analysis 2: Comparison: Low-Dose Ataluren vs Placebo; Analysis was performed using MMRM method including rank transformed 6MWD as the dependent variable; and rank transformed baseline 6MWD, treatment, visit, age (< 9 years vs. >= 9 years) and corticosteroid use (yes vs. no) stratification factors, and interaction between treatment and visit as independent variables; Test type: Other; p = 0.1490, Mixed Models Analysis; LS Mean Difference = 62.65, 95% CI 2-sided [-22.66 to 147.96], Standard Error of Mean 43.21

2. Secondary Outcome: Change From Baseline in Time to Stand From Supine Position at Week 48
Description: If the time taken to perform this test exceeded 30 seconds or if a participant could not perform this test due to disease progression, a value of 30 seconds was used. Change from baseline data has been reported.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
seconds
  Baseline | 12.25 (11.191) | 10.80 (9.924) | 11.50 (11.440)
  Change at Week 48: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48 | 3.00 (5.686) | 3.23 (5.761) | 3.24 (7.253)

3. Secondary Outcome: Change From Baseline in Time to Walk/Run 10 Meters at Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
seconds
  Baseline | 7.80 (5.243) | 7.45 (4.373) | 6.86 (2.813)
  Change at Week 48: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48 | 2.37 (6.149) | 1.68 (5.617) | 3.03 (6.691)

4. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs at Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
seconds
  Baseline | 7.63 (7.522) | 6.94 (6.474) | 6.04 (5.661)
  Change at Week 48: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48 | 3.51 (6.794) | 2.39 (4.618) | 4.79 (7.949)

5. Secondary Outcome: Change From Baseline in Time to Descend 4 Stairs at Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
seconds
  Baseline | 6.75 (7.219) | 6.08 (5.985) | 5.52 (5.753)
  Change at Week 48: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48 | 2.95 (7.323) | 2.41 (6.162) | 4.03 (7.828)

6. Secondary Outcome: Change From Baseline in Force Exerted During Knee Flexion and Extension, Elbow Flexion and Extension, and Shoulder Abduction at Week 48, as Assessed by Myometry
Description: Upper and lower extremity myometry was performed using a myometer following standardized procedures. Muscle groups evaluated included knee flexors, knee extensors, elbow flexors, elbow extensors, and shoulder abductors. Bilateral assessments were done and 3 measurements were recorded from each muscle group on each side if possible. Mean values for the left and right sides were calculated.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
pounds
  Baseline: Force during knee flexion | 12.45 (4.684) | 12.08 (4.217) | 11.06 (3.494)
  Change at Week 48: Force during knee flexion: number analyzed (Participants) | 59 | 57 | 55
  Change at Week 48: Force during knee flexion | 0.39 (3.148) | -0.07 (3.511) | 0.38 (2.991)
  Baseline: Force during knee extension: number analyzed (Participants) | 60 | 57 | 56
  Baseline: Force during knee extension | 12.71 (7.910) | 12.81 (5.753) | 12.96 (6.162)
  Change at Week 48: Force during knee extension: number analyzed (Participants) | 59 | 57 | 55
  Change at Week 48: Force during knee extension | -0.59 (3.511) | -0.63 (3.616) | -1.85 (3.899)
  Baseline: Force exerted during elbow flexion | 8.72 (4.709) | 7.66 (3.154) | 8.14 (2.972)
  Change at Week 48: Force during elbow flexion: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48: Force during elbow flexion | -0.50 (1.832) | -0.10 (1.680) | -0.35 (1.807)
  Baseline: Force during elbow extension | 6.81 (3.815) | 6.19 (3.083) | 6.77 (2.785)
  Change at Week 48: Force during elbow extension: number analyzed (Participants) | 59 | 57 | 56
  Change at Week 48: Force during elbow extension | -0.28 (1.473) | 0.10 (1.493) | -0.51 (2.333)

7. Secondary Outcome: Change From Baseline in Mean Activity Period/Day/Visit at Week 48, as Assessed by Step Activity Monitoring (SAM)
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean activity period/day/visit was computed for each participant. Mean obtained during Screening (Week -6 to -1) and following Week 1 visit were used as baseline data for analysis. For each day, an active period was defined as the first time after 3:00 AM that greater than (>) 2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was less than (<) 50 percent (%) of the mean active period across all days for that participant's visit.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
minutes
  Baseline: number analyzed (Participants) | 59 | 53 | 54
  Baseline | 756.84 (84.612) | 761.86 (76.984) | 751.71 (60.513)
  Change at Week 48: number analyzed (Participants) | 56 | 53 | 49
  Change at Week 48 | 0.87 (57.833) | -22.23 (84.759) | -19.91 (91.960)

8. Secondary Outcome: Change From Baseline in Mean Total Step Count/Day/Visit During the Active Periods at Week 48, as Assessed by SAM
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean total step count/day/visit during the active periods was computed for each participant. Mean obtained during Screening (Week -6 to -1) and following Week 1 visit were used as baseline data for analysis. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
steps/day
  Baseline: number analyzed (Participants) | 59 | 53 | 54
  Baseline | 5302.31 (1907.058) | 4870.13 (2165.522) | 5602.31 (2023.543)
  Change at Week 48: number analyzed (Participants) | 56 | 53 | 49
  Change at Week 48 | -615.14 (1468.452) | -676.46 (1717.535) | -908.34 (1999.969)

9. Secondary Outcome: Change From Baseline in Mean Total Step Count/Hour During the Active Period at Week 48, as Assessed by SAM
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean total step count/hour during the active periods for the days in a visit was computed for each participant. Mean obtained during Screening (Week -6 to -1) and following Week 1 visit were used as baseline data for analysis. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: steps/hour
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
steps/hour
  Baseline: number analyzed (Participants) | 59 | 53 | 54
  Baseline | 423.67 (168.754) | 383.62 (161.911) | 446.37 (160.666)
  Change at Week 48: number analyzed (Participants) | 56 | 53 | 49
  Change at Week 48 | -44.51 (125.154) | -42.23 (126.429) | -59.62 (153.054)

10. Secondary Outcome: Change From Baseline in Maximum Continuous 10-minute, 20-minute, 30-minute, and 60-minute Total Step Count at Week 48, as Assessed by SAM
Description: SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). The maximum continuous 10-minute, 20-minute, 30-minute, and 60-minute total step counts were computed for each participant. Mean obtained during Screening (Week -6 to -1) and following Week 1 visit were used as baseline data for analysis. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline, Week 48
Population: ITT population included all participants who were randomized and received any study treatment; and had a valid baseline, and at least one valid post-baseline 6MWD value. Here, 'Number analyzed' signifies participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
steps
  Baseline: 10-minute total step count: number analyzed (Participants) | 59 | 55 | 54
  Baseline: 10-minute total step count | 35.77 (10.222) | 32.24 (11.374) | 36.76 (8.935)
  Change at Week 48: 10-minute total step count: number analyzed (Participants) | 56 | 54 | 49
  Change at Week 48: 10-minute total step count | -2.77 (8.569) | -2.79 (6.355) | -3.97 (9.720)
  Baseline: 20-minute total step count: number analyzed (Participants) | 59 | 55 | 54
  Baseline: 20-minute total step count | 29.13 (9.272) | 25.68 (10.038) | 29.74 (8.205)
  Change at Week 48: 20-minute total step count: number analyzed (Participants) | 56 | 54 | 49
  Change at Week 48: 20-minute total step count | -2.49 (7.407) | -2.40 (5.806) | -3.55 (8.677)
  Baseline: 30-minute total step count: number analyzed (Participants) | 59 | 55 | 54
  Baseline: 30-minute total step count | 25.00 (8.053) | 22.08 (9.206) | 25.70 (7.350)
  Change at Week 48: 30-minute total step count: number analyzed (Participants) | 56 | 54 | 49
  Change at Week 48: 30-minute total step count | -2.08 (6.519) | -2.31 (5.505) | -3.03 (7.604)
  Baseline: 60-minute total step count: number analyzed (Participants) | 59 | 55 | 54
  Baseline: 60-minute total step count | 18.58 (6.210) | 16.52 (7.199) | 19.50 (5.887)
  Change at Week 48: 60-minute total step count: number analyzed (Participants) | 56 | 54 | 49
  Change at Week 48: 60-minute total step count | -1.50 (5.177) | -1.85 (4.616) | -2.33 (6.241)

11. Secondary Outcome: Change From Baseline in Percentage of Time During the Active Period Spent at Low Activity (Less Than or Equal to [≤] 15 Steps/Minute), Medium Activity (16-30 Steps/Minute), and High Activity (Greater Than [>]30 Steps/Minute) at Week 48
Description: SAM is a pedometer(worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again. Proportion of time during active periods spent at low activity(≤15 steps/minute), medium activity(16-30 steps/minute), and high activity(>30 steps/minute) were computed for each participant. Mean obtained during Screening and following Week 1 visit were used as baseline data for analysis. For each day, an active period was defined as first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline, Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
percentage of time
  Baseline: Time spent at low activity: number analyzed (Participants) | 59 | 53 | 54
  Baseline: Time spent at low activity | 32.91 (7.842) | 32.38 (8.213) | 32.86 (6.239)
  Change at Week 48: Time spent at low activity: number analyzed (Participants) | 56 | 53 | 49
  Change at Week 48: Time spent at low activity | -2.06 (7.903) | -1.12 (8.220) | -1.11 (5.586)
  Baseline: Time spent at medium activity: number analyzed (Participants) | 59 | 53 | 54
  Baseline: Time spent at medium activity | 11.11 (4.013) | 10.00 (3.656) | 11.84 (4.304)
  Change at Week 48: Time spent at medium activity: number analyzed (Participants) | 56 | 53 | 49
  Change at Week 48: Time spent at medium activity | -1.35 (3.348) | -0.69 (3.828) | -1.92 (4.178)
  Baseline: Time spent at high activity: number analyzed (Participants) | 59 | 53 | 54
  Baseline: Time spent at high activity | 6.59 (4.077) | 5.78 (3.785) | 7.17 (3.700)
  Change at Week 48: Time spent at high activity: number analyzed (Participants) | 54 | 52 | 48
  Change at Week 48: Time spent at high activity | -0.66 (2.790) | -0.96 (2.828) | -1.03 (3.783)

12. Secondary Outcome: Change From Baseline in Participant- Reported Health-Related Quality of Life (HRQL) as Measured by the Pediatric Quality of Life Inventory (PedsQL) Physical, Emotional, Social, and School Functioning Domain Scores at Week 48
Description: HRQL was measured via the PedsQL. The generic core module (including physical, emotional, social and school functioning scales) comprises 23 questions and the fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. The PedsQL was completed by both the participant and/or a parent/caregiver. Examples of items in each of the generic core module scales include: "It is hard for me to run"; "I feel sad or blue"; "I cannot do things that other kids my age can do;" and "It is hard to pay attention in class." Each of the generic core module items was scored on a 5-point likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating better health-related quality of life. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline, Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units on a scale
  Baseline: Physical functioning score: number analyzed (Participants) | 58 | 56 | 56
  Baseline: Physical functioning score | 63.63 (20.029) | 59.27 (22.782) | 61.87 (19.411)
  Change at Week 48: Physical functioning score: number analyzed (Participants) | 54 | 55 | 50
  Change at Week 48: Physical functioning score | -0.94 (19.125) | 2.37 (25.105) | -1.00 (24.022)
  Baseline: Emotional functioning score: number analyzed (Participants) | 58 | 55 | 56
  Baseline: Emotional functioning score | 73.92 (20.418) | 73.70 (20.223) | 70.13 (19.332)
  Change at Week 48: Emotional functioning score: number analyzed (Participants) | 54 | 54 | 50
  Change at Week 48: Emotional functioning score | 2.36 (16.742) | -1.83 (23.725) | 4.30 (22.315)
  Baseline: Social functioning score: number analyzed (Participants) | 58 | 55 | 55
  Baseline: Social functioning score | 67.50 (21.749) | 65.09 (18.421) | 63.36 (20.476)
  Change at Week 48: Social functioning score: number analyzed (Participants) | 54 | 54 | 51
  Change at Week 48: Social functioning score | 5.37 (20.463) | 3.89 (21.841) | 7.75 (18.870)
  Baseline: School functioning score: number analyzed (Participants) | 58 | 55 | 54
  Baseline: School functioning score | 67.72 (19.276) | 64.55 (20.396) | 64.65 (17.841)
  Change at Week 48: School functioning score: number analyzed (Participants) | 52 | 54 | 49
  Change at Week 48: School functioning score | 3.61 (13.008) | 6.11 (23.765) | 4.06 (23.244)

13. Secondary Outcome: Change From Baseline in Parent/Caregiver- Reported HRQL as Measured by the PedsQL Physical, Emotional, Social, and School Functioning Domain Scores at Week 48
Description: as for outcome 12
Time Frame: Baseline, Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units on a scale
  Baseline: Physical functioning score: number analyzed (Participants) | 60 | 56 | 57
  Baseline: Physical functioning score | 56.15 (19.955) | 54.96 (20.592) | 51.47 (19.274)
  Change at Week 48: Physical functioning score: number analyzed (Participants) | 59 | 56 | 57
  Change at Week 48: Physical functioning score | 0.03 (17.088) | -3.10 (16.550) | 0.23 (23.712)
  Baseline: Emotional functioning score: number analyzed (Participants) | 60 | 56 | 57
  Baseline: Emotional functioning score | 70.08 (16.836) | 69.11 (18.711) | 65.96 (17.964)
  Change at Week 48: Emotional functioning score: number analyzed (Participants) | 59 | 56 | 57
  Change at Week 48: Emotional functioning score | 4.07 (15.382) | 3.39 (18.068) | 1.21 (17.794)
  Baseline: Social functioning score: number analyzed (Participants) | 60 | 56 | 57
  Baseline: Social functioning score | 61.58 (15.825) | 62.77 (16.540) | 55.79 (18.269)
  Change at Week 48: Social functioning score: number analyzed (Participants) | 59 | 56 | 57
  Change at Week 48: Social functioning score | -0.40 (18.470) | -1.09 (14.268) | 3.71 (14.130)
  Baseline: School functioning score: number analyzed (Participants) | 60 | 56 | 57
  Baseline: School functioning score | 66.17 (18.258) | 66.16 (16.320) | 61.93 (13.587)
  Change at Week 48: School functioning score: number analyzed (Participants) | 58 | 56 | 56
  Change at Week 48: School functioning score | 2.73 (18.490) | -2.32 (15.462) | 3.48 (13.913)

14. Secondary Outcome: Change From Baseline in Participant-Reported HRQL as Measured by the Total Fatigue Scale Score at Week 48
Description: HRQL was measured via the PedsQL. The fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. PedsQL was completed by both the participant and/or a parent/caregiver. Fatigue-specific module obtains information relating to items such as: "I feel too tired to do things that I like to do"; "I spend a lot of time in bed"; and "I have trouble remembering more than one thing at a time;" Each of the fatigue-specific module items was scored on a 5-point likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating less fatigue. Total score was the sum of all items over the number of items answered on all scales. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units on a scale
  Baseline: number analyzed (Participants) | 58 | 55 | 54
  Baseline | 69.47 (16.525) | 71.62 (16.474) | 69.70 (15.263)
  Change at Week 48: number analyzed (Participants) | 55 | 54 | 52
  Change at Week 48 | 6.95 (13.460) | 0.45 (23.068) | 3.92 (16.512)

15. Secondary Outcome: Change From Baseline in Parent/Caregiver-Reported HRQL as Measured by the Total Fatigue Scale Score at Week 48
Description: HRQL was measured via the PedsQL. The fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. The PedsQL was completed by both the participant and/or a parent/caregiver. Fatigue-specific module obtains information relating to items such as: "I feel too tired to do things that I like to do"; "I spend a lot of time in bed"; and "I have trouble remembering more than one thing at a time;" Each of the fatigue-specific module items was scored on a 5-point likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating less fatigue. Total score was the sum of all items over the number of items answered on all scales. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units on a scale
  Baseline: number analyzed (Participants) | 60 | 56 | 57
  Baseline | 73.39 (13.671) | 70.71 (12.720) | 68.27 (13.170)
  Change at Week 48: number analyzed (Participants) | 58 | 54 | 57
  Change at Week 48 | 1.97 (13.873) | 1.27 (12.095) | 2.51 (12.039)

16. Secondary Outcome: Parent/Caregiver-Reported Treatment Satisfaction Questionnaire for Medication (TSQM) Score
Description: TSQM consisted of 14 questions about treatment satisfaction with drug in 4 domains: Effectiveness (Questions 1-3 scored as 1 [extremely dissatisfied] to 7 [extremely satisfied]), Side Effects (question 4 scored as 0 [no] or 1 [yes]; question 5 scored as 1 [extremely bothersome] to 5 [not at all bothersome]; questions 6 - 8 scored as 1 [a great deal] to 5 [not at all]), Convenience (questions 9 and 10 scored as 1 [extremely difficult] to 7 [extremely easy]; question 11 scored as 1 [extremely inconvenient] to 5 [extremely convenient]) and Global Satisfaction (question 12 scored as 1 [not at all confident] to 7 [extremely confident]; question 13 scored as 1 [not at all certain] to 5 [extremely certain]; question 14 scored as 1 [extremely dissatisfied] to 5 [extremely satisfied]). The scores of each of the domains were added together and an algorithm was used to create a score of 0 to 100, with higher scores indicating better treatment satisfaction.
Time Frame: Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units on a scale
  Effectiveness score: number analyzed (Participants) | 53 | 55 | 53
  Effectiveness score | 55.97 (27.796) | 54.60 (22.307) | 51.26 (23.536)
  Side-effects score: number analyzed (Participants) | 55 | 56 | 55
  Side-effects score | 96.36 (11.199) | 97.77 (7.578) | 96.89 (8.874)
  Convenience score: number analyzed (Participants) | 57 | 56 | 55
  Convenience score | 55.85 (17.008) | 58.23 (19.040) | 60.91 (16.665)
  Global satisfaction score: number analyzed (Participants) | 55 | 56 | 55
  Global satisfaction score | 61.04 (25.967) | 61.19 (23.691) | 57.56 (21.851)

17. Secondary Outcome: Change From Baseline in Participant/Caregiver-Reported Number of Daily Accidental Falls at Week 48
Description: Number of falls was determined by daily diary records maintained by participants and/or parent/caregivers.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: falls/day
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
falls/day
  Baseline: number analyzed (Participants) | 54 | 48 | 48
  Baseline | 0.40 (0.597) | 0.27 (0.480) | 0.54 (0.943)
  Change at Week 48: number analyzed (Participants) | 52 | 47 | 44
  Change at Week 48 | -0.10 (0.466) | -0.06 (0.501) | 0.20 (1.282)

18. Secondary Outcome: Change From Baseline in Number of Digits Recalled Forwards and Backwards on Digit Span Task at Week 48
Description: Basic attention and working memory was measured using the digit span task. A series of digits (0-9) were presented to the child in an auditory format only. The task had 2 parts; in the forward condition, the child was requested to repeat back the digits in the order they were presented and in the backward condition, he was requested to reverse the order of presentation. A raw score of the total number of correct responses was converted to an age-scaled-score (z-score) by subtracting the corresponding mean and dividing by the corresponding standard deviation of a reference population for that age.
Time Frame: Baseline, Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
z-score
  Baseline: Forward condition: number analyzed (Participants) | 59 | 56 | 55
  Baseline: Forward condition | 3.59 (2.554) | 2.89 (2.180) | 2.84 (1.675)
  Change at Week 48: Forward condition: number analyzed (Participants) | 57 | 54 | 52
  Change at Week 48: Forward condition | 0.39 (1.677) | 0.50 (1.767) | 0.40 (1.550)
  Baseline: Backward condition: number analyzed (Participants) | 59 | 56 | 54
  Baseline: Backward condition | 1.73 (1.846) | 1.70 (1.868) | 1.59 (1.460)
  Change at Week 48: Backward condition: number analyzed (Participants) | 57 | 54 | 51
  Change at Week 48: Backward condition | 0.56 (1.500) | 0.33 (1.441) | 0.59 (1.203)

19. Secondary Outcome: Change From Baseline in Heart Rate Before, During, and After Each 6MWT at Week 48, as Assessed by Heart Rate Monitoring With the Polar® RS400
Description: The heart rate was measured with a Polar RS400 heart rate monitor, which consists of a transmitter strap worn around the chest and a wristwatch receiver. The monitor produces a digital text file with 1 value per minute that represents the mean heart rate for that minute. Mean heart rates values were collected prior to, during, and after the 6MWT. The participant rested for 5 minutes in a sitting position prior to the 6MWT, and the mean heart rate for the last minute of this rest period was collected and documented as the resting heart rate. During the 6MWT, the mean heart rate was collected and documented as the active heart rate. After completing the 6MWT and resting for 3 minutes, the mean heart rate for 1 minute was collected and documented as the recovery heart rate.
Time Frame: Baseline, Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
beats/minute
  Baseline: Resting heart rate | 105.47 (12.908) | 109.70 (9.908) | 104.07 (11.588)
  Change at Week 48: Resting heart rate: number analyzed (Participants) | 54 | 53 | 50
  Change at Week 48: Resting heart rate | -0.63 (13.008) | -0.36 (10.223) | -0.26 (15.614)
  Baseline: Active heart rate: number analyzed (Participants) | 60 | 56 | 57
  Baseline: Active heart rate | 142.67 (18.070) | 141.77 (15.574) | 136.67 (20.713)
  Change at Week 48: Active heart rate: number analyzed (Participants) | 53 | 49 | 48
  Change at Week 48: Active heart rate | -5.00 (21.976) | 2.39 (19.095) | 1.65 (21.295)
  Baseline: Recovery heart rate: number analyzed (Participants) | 60 | 56 | 57
  Baseline: Recovery heart rate | 109.90 (12.633) | 113.48 (10.340) | 107.86 (12.066)
  Change at Week 48: Recovery heart rate: number analyzed (Participants) | 53 | 49 | 48
  Change at Week 48: Recovery heart rate | -0.23 (13.475) | -1.33 (13.270) | 0.54 (15.181)

20. Secondary Outcome: Change From Baseline in Serum Concentration of Creatine Kinase (CK) at Week 48
Description: Blood samples collected for chemistry assays were used to quantify serum CK concentrations. Serum CK was assessed as a potential biomarker for muscle fragility, with a reduction in serum CK considered to be a positive outcome.
Time Frame: Baseline, Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units/liter (U/L)
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
units/liter (U/L)
  Baseline | 10853.65 (6251.136) | 12084.70 (7772.631) | 10569.60 (6488.477)
  Change at Week 48: number analyzed (Participants) | 58 | 57 | 55
  Change at Week 48 | -1680.09 (4264.769) | -2146.32 (7151.944) | -1235.13 (4323.943)

21. Secondary Outcome: Percent Change From Pre-Treatment Visit (1 Week Prior to Baseline Visit) in Biceps Muscle Dystrophin Expression at Post-Treatment Visit (Week 36), as Determined by Immunofluorescence
Description: Immunofluorescence evidence of a change in dystrophin expression on biceps muscle biopsy was defined as an increase in the staining of the sarcolemmal membrane with an antibody to the C-terminal portion of the dystrophin protein (excluding revertant fibers) between the pre-treatment (1 week prior to Baseline visit) and post-treatment (Week 36) biopsies. The biceps muscle was biopsied from one arm for confirmation of the absence or reduced levels of dystrophin prior to treatment initiation and from the other arm to assess for production of dystrophin post-treatment.
Time Frame: Pre-Treatment (1 week prior to baseline), post-treatment (Week 36)
Population: As-treated population included all randomized participants who actually received any study treatment. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
percent change
  Pre-treatment: number analyzed (Participants) | 60 | 55 | 56
  Pre-treatment | 336.096 (138.9753) | 359.797 (142.7361) | 357.271 (139.6650)
  Percent change post-treatment: number analyzed (Participants) | 59 | 55 | 56
  Percent change post-treatment | -1.278 (27.7432) | -2.128 (28.8287) | -0.898 (19.2112)

22. Other Pre Specified Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. Treatment-emergent adverse event (TEAE) was defined as an adverse event that occurred or worsened in the period extending from first dose of study drug to 6 weeks after the last dose of study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 54
Population: As-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
percentage of participants | 95.0 | 96.5 | 98.2

23. Other Pre Specified Outcome: Study Drug Compliance
Description: Study drug compliance was assessed by participant daily diary and quantification of used and unused study drug. Compliance was assessed in terms of the percentage of drug actually taken relative to the amount that should have been taken during the study.
Time Frame: Baseline to Week 48
Population: As-treated population included all randomized participants who actually received any study treatment.
Measure: Median (Full Range); unit: percentage of drug
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Number analyzed (Participants) | 60 | 57 | 57
percentage of drug | 97.87 [34.9 to 99.6] | 97.03 [64.5 to 99.8] | 97.74 [76.6 to 99.9]

ADVERSE EVENTS:
Time Frame: Baseline up to 6 weeks after the last dose of study drug (Week 54)
Description: As-treated population included all randomized participants who actually received any study treatment.
Arm/Group | High-Dose Ataluren | Low-Dose Ataluren | Placebo
Serious Adverse Events (participants affected / at risk) | 2/60 | 2/57 | 3/57
Other Adverse Events (participants affected / at risk) | 58/60 | 56/57 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose Ataluren (N=60) | Low-Dose Ataluren (N=57) | Placebo (N=57)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Ataluren (N=60) | Low-Dose Ataluren (N=57) | Placebo (N=57)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dilatation ventricular (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Macroglossia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (3) | 3 (3)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 2 (2) | 2 (5) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelid cyst (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 12 (23) | 8 (8) | 4 (10)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 13 (32) | 9 (18) | 9 (13)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 2 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 18 (39) | 11 (15) | 15 (20)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 10 (10) | 5 (5) | 4 (4)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (16) | 8 (16) | 7 (9)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 5 (7) | 4 (4) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 28 (72) | 33 (88) | 22 (48)
Adhesion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (5) | 3 (4) | 2 (2)
Disease progression (General disorders) | 5 (5) | 4 (4) | 6 (6)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 2 (2) | 2 (3)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 4 (4) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 1 (4) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (10) | 14 (21) | 12 (14)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 4 (5) | 3 (4) | 4 (4)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (7) | 10 (10) | 4 (7)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 4 (4) | 3 (4)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 7 (9) | 6 (8) | 8 (9)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Measles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (15) | 13 (22) | 13 (17)
Oral candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
Paronychia (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 1 (3) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (4) | 7 (11) | 2 (2)
Roseola (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (7)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (4)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (18) | 9 (16) | 12 (17)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 3 (4) | 3 (3) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 8 (9) | 8 (10) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 4 (6)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (14) | 11 (15) | 7 (7)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 3 (3) | 6 (8) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 2 (2)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 11 (17) | 10 (13) | 10 (14)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood aldosterone increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Immunoglobulins decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Renin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Thyroxine free increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Thyroxine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine colour abnormal (Investigations) | 0 (0) | 1 (1) | 1 (3)
Weight decreased (Investigations) | 5 (5) | 6 (6) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 5 (6) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (15) | 9 (9) | 5 (10)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Joint contracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lordosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 5 (8)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (16) | 8 (12) | 6 (7)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Trendelenburg's symptom (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3) | 1 (1)
Areflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (4) | 4 (5)
Headache (Nervous system disorders) | 16 (85) | 23 (69) | 14 (25)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (2) | 2 (4) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (3) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Encopresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Enuresis (Renal and urinary disorders) | 3 (4) | 4 (4) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Myoglobinuria (Renal and urinary disorders) | 1 (1) | 1 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Residual urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Strangury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (27) | 9 (14) | 13 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 3 (6) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (8) | 5 (9)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (7) | 4 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 6 (8)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7) | 5 (6)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 5 (9) | 4 (8) | 4 (7)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (6) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.